CLINICAL TRIAL: NCT02879604
Title: Cost-utility Study of a Group of Compensatory Cognitive Remediation in Schizophrenia
Acronym: Grecco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); University Hospital, Clermont-Ferrand (Other); Assistance Publique - Hôpitaux de Paris (Other); Hôpital Louis Mourier (Other); Centre Hospitalier Charles Perrens, Bordeaux (Other Government); University Hospital, Strasbourg (Other); Hospital Center Alpes-Isère (Other); Hôpitaux à Bron (Other); Fondation FondaMental (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL15_0503
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia
Keywords: cognitive remediation, cost-effectiveness analysis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compensatory cognitive training (Experimental): Compensatory cognitive training
  Interventions: Other: Compensatory cognitive training
- usual treatment (Placebo Comparator): usual treatment for shizophrenai
  Interventions: Other: Usual

INTERVENTIONS:
Other: Compensatory cognitive training — In addition to the usual care, method of compensatory cognitive remediation
  Other Names: CCT
  Arms: Compensatory cognitive training
Other: Usual — Usual care
  Arms: usual treatment

SUMMARY:
Significant cognitive impairment (executive functions, memory, attention) is common in schizophrenia affecting up to 80% of patients. But pharmacological treatments (typical and atypical antipsychotic) do not have impact on cognitive functioning. For over 20 years, alternative non-pharmacological therapeutics have been developed in schizophrenia. These techniques called cognitive remediation specifically target cognitive deficits. The first cognitive remediation available for patients was designed to stimulate new learning, or relearning, of cognitive tasks, and thus to improve certain deficient domains. These procedures were efficient in improving cognition as measured by neurocognitive tests but their impact on functioning and daily life was weak. In a second time, compensatory remediation has been developed. Compensatory approaches seek to make improvements in the patient's functioning by avoiding areas of impairment and recruiting other intact cognitive domains or by creating a supportive external environment. In recent meta-analysis compensatory remediation has larger effect-size than classical cognitive remediation, with an impact on patients psychosocial functioning. Recently, Dr E. Twamley (University of California) developed and tested a group-based, manualized, compensatory cognitive training intervention.

Compensatory cognitive training (CCT) is a low-tech, brief intervention and is easily transposable in community care. Our team translated this method into French. The investigators planned a cost -utility study between CCT and treatment as usual in schizophrenia patients with less than 10 years of evolution.

DETAILED DESCRIPTION:
This study will take place over 3 years with a recruitment period of 18 months. After verification of the eligibility criteria and signature of the consent, the patients will be divided into 2 groups by randomization: the intervention group and the control group. The duration of participation of the subjects will be 12 months. Assessments are available in 4 steps (V1 at inclusion, V2 at 3 months, V3 at 6 months and V4 at 12 months). These visits include an assessment of the functioning of patients, symptomatology, quality of life, treatment and care received at all visits, occupational activity and cognitive assessment and social knowledge at V1 and V4.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic with schizophrénie
* Less than 10 years of the evolution of the disease

Exclusion Criteria:

* History of severe cranial trauma and / or neurological pathology with cognitive impairment
* Ongoing participation in another study for treatment of negative or cognitive symptoms
* Ongoing participation in a study on management in psychotherapy for cognitive disorders and negative symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Cost-utility questionnaire | 12 months
  Cost difference between the 2 group of patients

SECONDARY OUTCOMES:
Functioning questionnaire | 3 months
  FROGS, Functional Remission of General Schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Delphine DC CAPDEVIELLE, MD-PhD, Study Director — Montpellier University Hospital
Locations (9):
- France (9):
  - Charles Perrens Hospital, Bordeaux
  - Le Vinatier Hospital, Bron
  - Gabriel-Montpied Univesity Hospital, Clermont-Ferrand
  - Louis Mourier Hospital, Colombes
  - Chenevier Hospital, Créteil
  - La Conception Hospital, Marseille
  - Montpellier University Hospital, Montpellier
  - Alpes Isère Hospital, Saint-Égrève
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No